CLINICAL TRIAL: NCT05001230
Title: Retrospective Study on Sexual Health in the Aftermath of an Obstetric Lesion of the Anal Sphincter
Acronym: LOSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8296
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-08

CONDITIONS: Lesions of the Anal Sphincter
Keywords: Lesions of the anal sphincter; Anal sphincter; Sexual health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lesions of the anal sphincter complicate 0.8% of childbirth in France. The sexual health of patients following this type of lesion is little studied, there are only about twenty articles on the subject.

The objective of this search is to study of the obstetric lesions of the anal sphincter

ELIGIBILITY:
Inclusion criteria:

* Adult woman (≥18 years old)
* Patient who gave birth at term to a child born living in the maternity hospitals of Strasbourg University Hospital between 01/01/2019 and 12/31/2019
* Single pregnancy
* 3rd degree or 4th degree perineal tear
* Intact perineum (control group)
* Good understanding of French orally
* Patient accepting to participate in the satisfaction telephone interview and not having expressed her opposition to the reuse of her data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Cesarean delivery
* Multiple pregnancy
* Premature delivery
* stillborn child
* impossibility of providing the subject with enlightened information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or guardianship
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman who gave birth at term to a child born living in the maternity hospitals of Strasbourg University Hospital between 01/01/2019 and 12/31/2019
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of obstetric lesions of the anal sphincter | Files analysed retrospectively from January 01, 2019 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Solène PETRY, MD, Principal Investigator — Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France